CLINICAL TRIAL: NCT03525288
Title: PSMA-PET Guided Radiotherapy in Patients With High-Risk, Recurrent, or Oligometastatic Prostate Cancer
Brief Title: PSMA-PET Guided Radiotherapy
Acronym: PSMA-PETgRT
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17.229; PERA GU17.1 (Registry Identifier: PERA)
Record Dates: First submitted 2018-03-19; First posted 2018-05-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are randomly selected from a standard-care cohort.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSMA-PETgRT (Experimental): PSMA-PET/CT imaging is performed during treatment planning. Treating physicians are informed of test results and advised to include up to 5 PSMA-PET avid sites distant to the prostate gland, if present, in the radiotherapy treatment plan.
  Interventions: Radiation: PSMA -PET/CT simulation
- Standard (Active Comparator): Patient's receive standard care radiotherapy and do not undergo PSMA-PET/CT imaging.
  Interventions: Radiation: Standard-care simulation

INTERVENTIONS:
Radiation: PSMA -PET/CT simulation — * PET/CT simulation.
  * If no additional lesions detected: RT as planned per standard care.
  * If PSMA-PET/CT imaging consistent with oligometastases (1-5 lesions): all lesions must be treated with definitive RT.
  * If PSMA-PET/CT imaging consistent with widely metastatic disease (>5 lesions): treatment of all detected disease with RT is not recommended, but treatment of the primary site as initially planned is encouraged.
  Arms: PSMA-PETgRT
Radiation: Standard-care simulation — No PSMA-PET/CT as part of RT treatment planning.
  Arms: Standard

SUMMARY:
PSMA PET/CT has demonstrated higher sensitivity in detecting metastases than current imaging standard of care (CT and bone scan). [18F]DCFPyL is a promising high-sensitivity second generation PSMA-targeted urea-based PET probe. The hypothesis is that definitive radiotherapy (RT) informed by PSMA-PET findings will lead to improved cancer control outcomes compared to RT guided by conventional staging only. This study utilizes cmRCT design in companion to PERA (Partnership initiative for the Evaluation of technological innovation in Radiotherapy).

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in PERA (CHUM CER 17.0.32) and consented to contact for investigational trials.
2. Histological diagnosis of prostate cancer planned for curative-intent radiotherapy.
3. ECOG 0-1
4. Charlson Cormobidity Index ≤ 4
5. High-risk of distant metastases as defined by any of:

   1. Oligometastases (≤5) (regional or distant) identified on conventional staging, with ≤ 3 metastasis in any non-bone organ. For a spine metastasis, direct involvement of adjacent spinal segments would still be considered as "one" tumour. For nodal metastases, more than one involved lymph node in the same ipsilateral nodal region/chain would still count as "one" tumour. Defined nodal regions for this protocol include inguinal, external iliac, internal iliac, common iliac, retroperitoneal, hilar/mediastinal, anterior cervical, posterior cervical, and axillary. Metastases in all other organs that are within 1cm of each other will be considered as "one" tumour.
   2. Subjects with newly diagnosed high-risk (NCCN) localized prostate cancer and CAPRA score 6-10.
   3. Subjects with a prior history of treated prostate cancer (RP or RT), and biochemical failure (Phoenix-RT or>0.2ng/ml-RP)
6. Standard staging (bone scan, CT pelvis) within 12 weeks of consent.

Exclusion Criteria:

1. Prior androgen deprivation therapy terminated < 12 months prior to enrollment.
2. Prior or planned PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 5 years
  Time to failure event

SECONDARY OUTCOMES:
Acute and delayed toxicities | 5 years
  Rate of Attributable Gr2+ toxicities (CTCAE v4.0)
Rate of failure | 5 years
  Event rates
Survival | 5 years
  Event rates
Health-related quality of life | 5 years
  Qol measures
Detection yield of PSMA PET imaging | 2 years
  Rate of new lesions identified on imaging

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - CSSSL - Cité de la Santé Laval, Laval, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU de Québec, Québec, Quebec

REFERENCES:
- [Derived] Belliveau C, Saad F, Duplan D, Petit C, Delouya G, Taussky D, Barkati M, Lambert C, Beauchemin MC, Clavel S, Mok G, Igidbashian L, Gauthier-Pare AS, Nguyen TV, McLaughlin PY, Keu KV, DaSilva JN, Juneau D, Menard C. Prostate-Specific Membrane Antigen PET-Guided Intensification of Salvage Radiotherapy After Radical Prostatectomy: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2025 Oct 2:e253746. doi: 10.1001/jamaoncol.2025.3746. Online ahead of print. PMID 41037308
- [Derived] Petit C, Delouya G, Taussky D, Barkati M, Lambert C, Beauchemin MC, Clavel S, Mok G, Pare AG, Nguyen TV, Duplan D, Keu KV, Saad F, Juneau D, Menard C. PSMA-PET/CT-Guided Intensification of Radiation Therapy for Prostate Cancer (PSMAgRT): Findings of Detection Rate, Effect on Cancer Management, and Early Toxicity From a Phase 2 Randomized Controlled Trial. Int J Radiat Oncol Biol Phys. 2023 Jul 15;116(4):779-787. doi: 10.1016/j.ijrobp.2022.12.055. Epub 2023 Jan 11. PMID 36639035